CLINICAL TRIAL: NCT03509363
Title: Comparisons Between the Effectiveness of Mobile Video-guided and Paper-based Home Exercise Programs on Improving Exercise Adherence, Self-Efficacy for Exercise and Functional Outcomes of Patients With Stroke a Single-blind Randomized Controlled Trial
Brief Title: Pilot Study on Comparisons Between the Effectiveness of Mobile Video-guided and Paper-based Home Exercise Programs of Patients With Stroke Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tai Po Hospital (Other Government)
Collaborators: Shatin Hospital (Other)
Responsible Party: Principal Investigator, Bryan Ping Ho CHUNG, Principal Investigator, Tai Po Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TPH-PT-001
Record Dates: First submitted 2018-04-17; First posted 2018-04-26 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: randomized, controlled
Who Masked: Outcomes Assessor
Masking Description: All research study personnel, including those who collect data and assess outcomes will be blinded to the group assignment. The envelopes and the randomization list will not be revealed to any of the study personnel until completion of recruitment and data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants allocated to the intervention group will be prescribed a set of exercise video with QR code provided in home exercise pamphlets and they have to perform the prescribed exercises under the guidance of video.The content of home exercise program in both groups is the same and is based on the recommendations from the National Stroke Foundation Clinical Guidelines, including mobilization exercise, strengthening exercise and balance training which is tailor-made for different mobility level of stroke patients. Suitability of participating home exercise program will be assessed by physiotherapists based on environmental risk, fall risk and competence of patients or carers in performing exercise with patients. The number of exercises prescribed, frequency and intensity of exercise varies from participants and will be determinated by physiotherapists
  Interventions: Behavioral: Stroke physiotherapy home exercise video
- Control (No Intervention): Participants in control group will be given instructions for their home exercise program in a traditional pamphlet includes photographs and instructions of exercise demonstration.

INTERVENTIONS:
Behavioral: Stroke physiotherapy home exercise video — a set of exercise video with QR code provided in home exercise pamphlets
  Other Names: exercise video
  Arms: Intervention

SUMMARY:
This is a pilot study and a randomized, controlled, assessor-blinded clinical trial for patients who will complete the inpatient Stroke Rehabilitation Program in the Department of Medical and Geriatrics of Tai Po Hospital and Shatin Hospital from June 2018 to March 2019. The objective of the study is to compare the effectiveness of video-guided exercise program and standard paperbased home exercise program on adherence of exercise, self-efficacy and improving functional outcomes in patients with stroke within 3-month follow-up.

DETAILED DESCRIPTION:
In Hong Kong, stroke patients would be referred to ambulatory services, such as geriatric day hospital, or domestic physiotherapy service to continue their stroke rehabilitation after discharge from hospital care. However, some patients could not attend ambulatory services due to vary difficulties, such as transportation and absence of carers. The low frequency of domestic physiotherapy service also reduced the effectiveness of rehabilitation of patients. Traditionally, for continuation of training at home, therapists would prescribe home exercises programs in paper-based format to stroke patients prior to discharge. However, evidence showed that written and pictorial home exercise prescription does not lead to better adherence to a home exercise programme compared to having no written and pictorial instructions for patients with stroke less than 4 months. It was suggested that the barriers to adherence of home exercise including low self-efficacy and delivery mode of training program. It is worthwhile for physiotherapists to investigate the mode of delivery to enhance exercise adherence and selfefficacy of post-discharge home exercise for patients with stroke. Recent survey concerning the development of smart technology revealed that 80% of global internet users owned a smart phone and 47% owned a tablet. Thus, the increasing accessibility of smart technology offers an opportunity to advance the mode of delivery of exercise program so as to benefit patients of stroke from increase the adherence and self-efficacy of home exercises. The evidences of using smart technology to enhance adherence of home exercise have reported inconsistent results. A study showed that home exercise programmes filmed on an electronic tablet, with an automated reminder, was not superior to standard paper-based home exercise programmes in terms of adherence, motor function, or satisfaction for patients recovering from stroke. In contrast, another study showed that people with musculoskeletal conditions adhere better to their home exercise programs when the programs are provided on an app with remote support compared to paper handouts; although the clinical importance of this added adherence is unclear. This is a pilot study and a randomized, controlled, assessor-blinded clinical trial for patients who will complete the inpatient Stroke Rehabilitation Program in the Department of Medical and Geriatrics of Tai Po Hospital and Shatin Hospital from June 2018 to March 2019. The objective of the study is to compare the effectiveness of video-guided exercise program and standard paperbased home exercise program on adherence of exercise, self-efficacy and improving functional outcomes in patients with stroke within 3-month follow-up. Eligible subjects will then be randomly assigned to either Intervention Group or Control Group in a 1:1 ratio.

Investigators who are responsible for data collection will be blinded to the group allocation. Pre-discharge training sessions last for 10- 15 minutes will be provided to patients, and their carers if any, of both groups in order to make them familiar with the selected home exercises and the technique of using mobile phone to scan QR for intervention group. Participants allocated to the intervention group will be prescribed a set of exercise video with QR code provided in home exercise pamphlets and they have to perform the prescribed exercises under the guidance of video. On the other hand, participants in control group will be given instructions for their home exercise program in a traditional pamphlet includes photographs and instructions of exercise demonstration. The content of home exercise program in both groups is the same and is based on the recommendations from the National Stroke Foundation Clinical Guidelines, including mobilization exercise, strengthening exercise and balance training which is tailor-made for different mobility level of stroke patients. Suitability of participating home exercise program will be assessed by physiotherapists based on environmental risk, fall risk and competence of patients or carers in performing exercise with patients. The number of exercises prescribed, frequency and intensity of exercise varies from participants and will be determinated by physiotherapists. Outcome measures including self-reported exercise adherence, self-efficacy for exercise, Modified Functional Ambulatory Category and Modified Barthel Index will be assessed at 1 day, 1 month and 3 month after discharged on phone follow-up basis by a blinded-assessor. We aim to recruit 28 participants in each group.

ELIGIBILITY:
Inclusion Criteria:

* 1. Stroke as principle diagnosis. 2. Could follow gesture and instructions of exercise training. 3. Could sit independently without back support for 2 minutes (MFAC Category II Sitter).

  4. Discharged home without any further training in ambulatory service such as Geriatric Day Hospital (GDH) and domestic physiotherapy services.

  5. Participants or their carers have smart devices such as smart phones or tablets that are able to scan QR code and connect to the Internet.

  6. Participants or carers could read Chinese.

Exclusion Criteria:

* 1. Participants who could walk independently with or without walking aids (MFAC Category 6, 7) before discharge from Tai Po Hospital and Shatin Hospital medical unit.

  2. Participants and their carers have visual or cognitive impairments that would prevent use of smart devices.

  3. Medical condition unstable

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Chinese version of the Modified Barthel Index | 3 months
  MBI was used to assess patients' basic activities of daily living (ADL) in this study. MBI measures the participant's performance on ten functional items including self-care, continence, and locomotion.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Ho CHUNG, MSc, Principal Investigator — Hospital Authority, Hong Kong
Locations (1):
- Tai Po Hospital, Hong Kong, Hong Kong